CLINICAL TRIAL: NCT03835728
Title: Exploratory Study of Efficacy of Ocrelizumab in Autoimmune Encephalitis
Brief Title: Efficacy of Ocrelizumab in Autoimmune Encephalitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failed to meet target enrollment and study was discontinued
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Steven Vernino, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2018-0185
Record Dates: First submitted 2019-02-05; First posted 2019-02-11 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System | interventions — ocrelizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Active Comparator): Ocrelizumab will be administered 3 times over a 1 year study period. Subjects will receive a dose of 300 mg at week 0 (baseline) and again at week 2. The final dose of 600 mg will be administered at week 24.
  Interventions: Drug: Ocrelizumab
- Treatment Placebo Arm (Placebo Comparator): Saline will be used as the matching placebo
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ocrelizumab — Subjects will be randomized in a 1:1 fashion to receive infusion of Ocrelizumab (2 doses at 300 mg and 1 dose at 600 mg) or matched placebo. The 2 300 mg doses will be administered at day 2 and day 14. The 600 mg dose will be administered during the 6 month visit. The drug will be administered via infusion three times throughout the trial period: after the initial screening, at two weeks from initial infusion, and at 6 months.
  Arms: Treatment Arm
Drug: Saline — This will be the matching placebo used in the study.
  Arms: Treatment Placebo Arm

SUMMARY:
This pilot study is a randomized, double-blind, placebo controlled study of the efficacy of ocrelizumab in autoimmune encephalitis. Subjects with new diagnosis of autoimmune encephalitis will be invited to enroll in this study. Subjects will be randomized to receive ocrelizumab (an anti-CD20 therapy) or matched placebo, and will undergo three infusions over a six month period. Subjects will complete clinical visits over the study period, during which safety monitoring and neuropsychological assessments will be performed to assess for signs of clinical worsening from encephalitis. The primary outcome of this study is the proportion of patients who fail to complete the twelve month period without clinical worsening, as defined by the protocol. Subjects who experience early clinical worsening during the study may be offered open-label treatment with ocrelizumab at the discretion of the investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or greater
2. Able to obtain informed consent from patient or appropriate designee
3. Possible autoimmune encephalitis as defined by Table 1:

   1. Reasonable exclusion of alternative causes
   2. Subacute onset (< 3 months) of memory deficits, altered consciousness, and/or psychiatric symptoms
   3. One or more of the following:

      * CSF (cerebrospinal fluid) pleocytosis (>5 cells/µl corrected, if necessary, for traumatic lumbar puncture)
      * EEG (electroencephalogram) with epileptiform or focal slow wave abnormalities involving temporal lobes
      * Brain abnormalities on T2/FLAIR MRI restricted to the mesial temporal (limbic) lobes
      * Associated dyskinesias (faciobrachial dystonic movements or orofacial dyskinesias)
4. Completed initial treatment with iv steroids (at least 3000mg solumedrol) and plasma exchange (at least 3 exchanges) within the past 8 weeks
5. Presence of one (or more) of the following autoantibodies in serum or CSF

   * NMDA receptor
   * LGI1
   * CASPR2
   * DPPX

Exclusion Criteria:

1. Prior immunosuppression treatment in past year (other than steroids, intravenous immunoglobulin and plasma exchange)
2. Active malignancy requiring chemotherapy
3. Pregnancy
4. Evidence of active hepatitis or tuberculosis infection
5. Medical condition that (in investigators opinion) precludes the use of ocrelizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Vernino, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Graus F, Titulaer MJ, Balu R, Benseler S, Bien CG, Cellucci T, Cortese I, Dale RC, Gelfand JM, Geschwind M, Glaser CA, Honnorat J, Hoftberger R, Iizuka T, Irani SR, Lancaster E, Leypoldt F, Pruss H, Rae-Grant A, Reindl M, Rosenfeld MR, Rostasy K, Saiz A, Venkatesan A, Vincent A, Wandinger KP, Waters P, Dalmau J. A clinical approach to diagnosis of autoimmune encephalitis. Lancet Neurol. 2016 Apr;15(4):391-404. doi: 10.1016/S1474-4422(15)00401-9. Epub 2016 Feb 20. PMID 26906964
- [Background] Titulaer MJ, McCracken L, Gabilondo I, Armangue T, Glaser C, Iizuka T, Honig LS, Benseler SM, Kawachi I, Martinez-Hernandez E, Aguilar E, Gresa-Arribas N, Ryan-Florance N, Torrents A, Saiz A, Rosenfeld MR, Balice-Gordon R, Graus F, Dalmau J. Treatment and prognostic factors for long-term outcome in patients with anti-NMDA receptor encephalitis: an observational cohort study. Lancet Neurol. 2013 Feb;12(2):157-65. doi: 10.1016/S1474-4422(12)70310-1. Epub 2013 Jan 3. PMID 23290630
- [Background] Dubey D, Sawhney A, Greenberg B, Lowden A, Warnack W, Khemani P, Stuve O, Vernino S. The spectrum of autoimmune encephalopathies. J Neuroimmunol. 2015 Oct 15;287:93-7. doi: 10.1016/j.jneuroim.2015.08.014. Epub 2015 Aug 28. PMID 26439968
- [Derived] Blackburn KM, Denney DA, Hopkins SC, Vernino SA. Low Recruitment in a Double-Blind, Placebo-Controlled Trial of Ocrelizumab for Autoimmune Encephalitis: A Case Series and Review of Lessons Learned. Neurol Ther. 2022 Jun;11(2):893-903. doi: 10.1007/s40120-022-00327-x. Epub 2022 Feb 7. PMID 35129803

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Failed to meet target enrollment and study was discontinued
Period: Overall Study
Arm/Group | Treatment Arm | Treatment Placebo Arm
Started | 2 | 1
Completed (Completed is defined as completing study procedures according to protocol even if the participant met primary endpoint and discontinued prior to 12 months.) | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Treatment Placebo Arm | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Customized [Median (Full Range); unit: years]
  Age | 47.5 [25 to 70] | 44 [44 to 44] | 44 [25 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3
Encephalitis antibody [Count of Participants; unit: Participants]
  NMDAR Ab | 1 | 1 | 2
  LGI1 Ab | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Clinical Worsening
Description: The number of participants who had clinical worsening within 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Treatment Placebo Arm
Number analyzed (Participants) | 2 | 1
Participants | 0 | 1

2. Secondary Outcome: Time to Treatment Failure
Description: Definition of clinical worsening (treatment failure):
  1. Clinician or patient/caregiver perception of clinical decline
  2. Worsening of patient/family reported IADL (by one point or more)
  3. One of the following additional features:
     * Significant worsening of Texas Functional Living Scale (by ≥ 5 T points, 0.5 st deviation)
     * Other clinical worsening leading to hospitalization
Time Frame: 12 months
Population: There were no treatment failures in the treatment arm. Thus, there was no data for this secondary outcome measure in the treatment arm
Measure: Number; unit: weeks
Arm/Group | Treatment Arm | Treatment Placebo Arm
Number analyzed (Participants) | 0 | 1
weeks |  | 12

3. Secondary Outcome: Change in TFLS T-score (Texas Functional Living Scale) Score at 6 Months
Description: Change in TFLS T-score (Texas Functional Living Scale) scores at 6 months compared to baseline. - A performance-based measure of functional competence designed to assess instrumental activities of daily living (e.g., managing money) that are thought to be more susceptible to cognitive change than basic activities of daily living (e.g., dressing).
  Content and Structure: The TFLS is comprised of 24 items divided into four subscales assessing abilities related to Time, Money and Calculation, Communication, and Memory. Many items provide a range of possible points allowing the instrument to account for the varying levels of functioning that may be observed in clinical populations.
  Total raw score ranges between 0 and 50 with standardized T-score values between 20 and 66. The higher the score, the better the performance.
  Change in TFLS T-score was used in this study
Time Frame: Baseline, 6 month
Population: Participant in placebo arm met study endpoint prior to 6 month outcome measure so change in TFLS score at 6 months was not analyzable for efficacy purposes.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment Arm | Treatment Placebo Arm
Number analyzed (Participants) | 2 | 0
score on a scale | 12.75 [3 to 22.5] |

4. Secondary Outcome: Change in TFLS T Score (Texas Functional Living Scale) Score at 12 Months
Description: Change in TFLS T-score (Texas Functional Living Scale) scores at 12 months compared to baseline. - A performance-based measure of functional competence designed to assess instrumental activities of daily living (e.g., managing money) that are thought to be more susceptible to cognitive change than basic activities of daily living (e.g., dressing).
  Content and Structure: The TFLS is comprised of 24 items divided into four subscales assessing abilities related to Time, Money and Calculation, Communication, and Memory. Many items provide a range of possible points allowing the instrument to account for the varying levels of functioning that may be observed in clinical populations.
  Total raw score ranges between 0 and 50 with standardized T-score values between 20 and 66. The higher the score, the better the performance.
  Change in TFLS T-score was used in this study
Time Frame: Baseline, 12 months
Population: Participant in placebo arm met study endpoint prior to 6 month outcome measure so change in TFLS score at 12 months was not analyzable for efficacy purposes.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment Arm | Treatment Placebo Arm
Number analyzed (Participants) | 2 | 0
score on a scale | 24.5 [3 to 46] |

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment Arm | Treatment Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=2) | Treatment Placebo Arm (N=1)
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Elevated transaminases (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seizures (Nervous system disorders) | 2 (2) | 0 (0) — related to encephalitis - unrelated to treatment

LIMITATIONS AND CAVEATS:
Early termination of trial due to inadequate recruitment. Small numbers of subjects prevents definitive analysis of results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT03835728/Prot_SAP_000.pdf